Official Title: Addressing Tobacco in Public Housing Residents Identifiers: NCT03620708

Document Date: September 27, 2019

#### Statistical Analysis Plan

To assess for differences in outcomes between groups we will use chi-square for dichotomous outcomes and analysis of variance / analysis of covariance for continuous outcomes. We will consider covariates based on theoretical grounds (e.g., baseline cigarettes per day, baseline motivation to quit, financial disadvantage) and significant differences between groups at baseline. Significant results will be probed using Dunnett's method, whereby our comparison of interest was between the treatment conditions and control condition. We will further report effect size estimates (i.e., f for ANOVA; Cramer's V for chi-square) to help elucidate aspects of the pilot study that may be most beneficial. Data will also be examined based on the assumption of 'missing equals smoking' and carrying the last observation (i.e., baseline data) forward, as a relatively conservative means of handling data for the n=5 participants lost to follow-up. We will refer to additional analyses of imputed data as intent-to=treat (ITT) analyses.

## Outcome 1: A self-described "serious" attempt to quit smoking cigarettes since the initial study appointment, measured by the "Quitting Preparation and Actions Questionnaire."

We will use chi-square analysis to examine differences in proportion of the participants randomized to receive the three intervention groups with respect to making a serious quit attempt between the initial appointment and the 1-month follow-up period.

# Outcome 2: Self-reported contact with one of two treatment referrals provided at intervention since the time of the initial study appointment

We will use chi-square analysis to examine differences in proportion of the participants randomized to receive the three intervention groups with respect to seeking treatment at either the NJ QuitLine or a NJ Quitcenter (local tobacco dependence treatment clinic) between the initial appointment and the 1-month follow-up period.

#### Outcome 3: Self-reported cigarettes smoked per day

We will use Analysis of Covariance (ANCOVA) to examine differences in cigarettes smoked per day at the 1-month follow-up between participants randomized to the three intervention groups. Baseline cigarettes smoked per day and measures of motivation to quit will be included as covariates.

### Outcome 4: Motivation and Self-efficacy for quitting smoking measured via Importance, Confidence, & Readiness Questionnaire" (rated on a 0 to 10 scale)

We will use separate Analysis of Covariance (ANCOVA) to examine differences in a) Self-reported Importance of quitting, b) Self-reported Confidence in one's ability to qut, and c) Self-reported Readiness to quit at the 1-month follow-up between participants randomized to the three intervention groups. Baseline ratings of motivation to quit will be included as a covariates.

# Outcome 5: "Readiness to Quit Ladder" (with 10 non-numbered choices reflecting varying degrees of readiness

We will use Analysis of Covariance (ANCOVA) to examine differences in cigarettes smoked per day at the 1-month follow-up between participants randomized to the three intervention groups. Baseline score on the Readiness to Quit Ladder will be included as a covariate.